CLINICAL TRIAL: NCT01074671
Title: Colvin-Galloway Future® Annuloplasty Ring/Band Clinical Trial: Interventional Multi-center Prospective Clinical Outcome Study
Brief Title: CG Future® Annuloplasty Ring/Band Clinical Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Organization: Medtronic Cardiovascular (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRC-CS-2009-06
Record Dates: First submitted 2010-01-26; First posted 2010-02-24 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Mitral Valve Insufficiency
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- No control arm (Other): There is no control arm as part of the study design.
  Interventions: Device: CG Future Annuloplasty Ring/Band

INTERVENTIONS:
Device: CG Future Annuloplasty Ring/Band — A CG Future Annuloplasty Ring or Band will be implanted, following standard care
  Other Names: Colvin Galloway Future Annuloplasty Ring; Colvin Galloway Future Annuloplasty Band; CG Future Annuloplasty Ring; CG Future Annuloplasty Band

SUMMARY:
The primary goal of the study is to document the number of patients that are successfully implanted and benefit from the implantation of both a CG Future Annuloplasty ring or a band.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated the Patient Informed Consent (PIC);
* Indicated to have a surgical repair for a given degree of moderate to severe mitral valve regurgitation;
* Willing to return to the implanting hospital for a 9 month follow-up visit

Exclusion Criteria:

* Unwilling or inability to sign the PIC;
* Already participating in another investigational device study, if this would create bias and jeopardize scientific appropriate assessment of the current study endpoints;
* Life expectancy of less than one year;
* Pregnant or desire to be pregnant within 12 months of the study treatment;
* Less than 18 years and more than 85 years of age.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2009-06; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Identification of the patient population for which a CG Future Annuloplasty Ring or Band is chosen to repair the mitral valve insufficiency | Within 3 months prior to implantation
The percentage of patients that are chronically relieved from mitral valve insufficiency | Within 3 months prior to implantation and at 9 month follow-up
The level of mitral valve regurgitation | Within 3 months prior to implantation and at 9 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: D C Iliopoulos, Prof, Principal Investigator — Athens Medical Center, Greece; M Hendrikx, Dr, Principal Investigator — Virga Jesse Hospital, Hasselt, Belgium; K François, Dr, Principal Investigator — UZ Gent, Belgium; G El Khoury, Dr, Principal Investigator — Cliniques Universitaires Saint Luc, Brussels, Belgium; K Widenka, Dr, Principal Investigator — Szpital Wojewódzki Nr 2 w Rzeszowie, Poland; R. Haaverstad, Prof., Principal Investigator — Haukeland Universitetssykehus, Bergen, Norway; K Matschke, Dr., Principal Investigator — Technische Universitat Dresden, Germany; F Riess, Dr., Principal Investigator — Albertinen Krankenhaus Hamburg, Germany
Locations (8):
- Belgium (3):
  - Cliniques Universitaires Saint Luc, Brussels
  - UZ Gent, Ghent
  - Virga Jesse Hospital, Hasselt
- Germany (2):
  - Technische Universitat Dresden, Dresden
  - Albertinen Krankenhaus Hamburg, Hamburg
- Athens Medical Center, Athens, Greece
- Haukeland Universitetssykehus, Bergen, Norway
- Szpital Wojewódzki Nr 2 w Rzeszowie, Rzeszów, Poland

REFERENCES:
- See also: Related Info — http://www.medtronic.com